CLINICAL TRIAL: NCT05172973
Title: Safety and Effectiveness of Balloon-Expandable Bioprosthetic SAPIEN X4 Transcatheter Heart Valve in Failing Aortic Bioprosthetic Valves
Brief Title: ALLIANCE AVIV: Safety and Effectiveness of the SAPIEN X4 Transcatheter Heart Valve in Failing Aortic Bioprosthetic Valves
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05-AVIV
Record Dates: First submitted 2021-12-14; First posted 2021-12-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement (TAVR); Transcatheter aortic valve implantation (TAVI); SAPIEN X4; Valve-in-valve
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcatheter Aortic Valve Replacement (TAVR) - Surgical Valve (Experimental): TAVR implant in subjects with a failing aortic surgical valve.
  Interventions: Device: SAPIEN X4 THV
- Transcatheter Aortic Valve Replacement (TAVR) - THV (Experimental): TAVR implant in subjects with a failing aortic transcatheter heart valve (THV).
  Interventions: Device: SAPIEN X4 THV

INTERVENTIONS:
Device: SAPIEN X4 THV — Implantation of the SAPIEN X4 valve

SUMMARY:
The objective of this study is to establish the safety and effectiveness of the Edwards SAPIEN X4 Transcatheter Heart Valve (THV) in subjects who are at high or greater risk with a failing aortic bioprosthetic valve.

DETAILED DESCRIPTION:
Prospective, single arm, multicenter study

ELIGIBILITY:
Inclusion Criteria:

1. Failing aortic bioprosthetic valve demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency
2. Bioprosthetic valve size suitable for SAPIEN X4 THV
3. NYHA functional class ≥ II
4. Heart Team agrees the subject is at high or greater surgical risk
5. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Anatomical characteristics that would preclude safe femoral placement of the introducer sheath or safe passage of the delivery system
2. Failing valve has moderate or severe paravalvular regurgitation
3. Failing valve is unstable, rocking, or not structurally intact
4. Known severe patient-prosthesis mismatch or bioprosthetic valve with residual mean gradient > 20 mmHg at the end of the index procedure for implantation of the original valve
5. Increased risk of THV embolization
6. Surgical or transcatheter valve in the mitral position
7. Severe mitral regurgitation (> 3+) or ≥ moderate mitral stenosis
8. Need for mitral, tricuspid or pulmonic valve intervention within the next 12 months
9. Left ventricular ejection fraction < 20%
10. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
11. Increased risk of coronary artery obstruction after THV implantation
12. Myocardial infarction within 30 days prior to the study procedure
13. Hypertrophic cardiomyopathy with subvalvular obstruction
14. Subjects with planned concomitant ablation for atrial fibrillation
15. Clinically significant coronary artery disease requiring revascularization
16. Any surgical or transcatheter procedure within 30 days prior to the study procedure. Implantation of a permanent pacemaker or implantable cardioverter defibrillator is not considered an exclusion.
17. Any planned surgical or transcatheter intervention to be performed within 30 days following the study procedure
18. Endocarditis within 180 days prior to the study procedure
19. Stroke, transient ischemic attack or neurological signs and symptoms attributed to carotid or vertebrobasilar disease within 90 days prior to the study procedure
20. Hemodynamic or respiratory instability requiring inotropic or mechanical support within 30 days prior to the study procedure
21. Renal insufficiency and/or renal replacement therapy
22. Leukopenia, anemia, thrombocytopenia
23. Inability to tolerate or condition precluding treatment with antithrombotic therapy
24. Hypercoagulable state or other condition that increases risk of thrombosis
25. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with premedication
26. Subject refuses blood products
27. Body mass index > 50 kg/m2
28. Estimated life expectancy < 24 months
29. Female who is pregnant or lactating
30. Active SARS-CoV-2 infection or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
31. Participating in another investigational drug or device study that has not reached its primary endpoint
32. Subject considered to be part of a vulnerable population

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Non-hierarchical composite of death and stroke | 1 year
  The number of patients that died or had a stroke

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 30 days
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
KCCQ score | 1 year
New York Heart Association (NYHA) functional class | 30 days
  NYHA is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.
NYHA functional class | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Yadav, MD, Principal Investigator — Piedmont Atlanta Hospital; Robert Cubbedu, MD, Principal Investigator — Naples Community Hospital
Locations (35):
- United States (32):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Bay Area Structural Heart at Sutter Health, San Francisco, California
  - Kaiser San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - UC Health Medical Center of the Rockies, Loveland, Colorado
  - Naples Community Hospital Healthcare System, Naples, Florida
  - Emory University Atlanta, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University Chicago, Evanston, Illinois
  - Alexian Brothers Hospital Network, Lisle, Illinois
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital Detroit, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System Morristown, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - University of Buffalo, Buffalo, New York
  - Cornelll University New York, New York, New York
  - Columbia University Medical Center / NYPH, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Carolinas Health System, Charlotte, North Carolina
  - Novant Health and Vascular Institute, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Saint Thomas Health, Nashville, Tennessee
  - University of Texas Memorial Hermann, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Washington Seattle, Seattle, Washington
- Canada (3):
  - St. Paul's Hospital Vancouver, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- Universite Laval, Québec

IPD SHARING:
Plan to Share IPD: No